CLINICAL TRIAL: NCT06463548
Title: Clinical Study of Irinotecan Hydrochloride Liposome Injection Combined With Capecitabine and Lenvatinib for Second-line Treatment in Patients With Advanced or Metastatic Biliary Tract Carcinoma
Brief Title: Irinotecan Hydrochloride Liposome Combined With Capecitabine and Lenvatinib in Patients With Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunpeng Liu (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yunpeng Liu, Director, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-BTC-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Capecitabine; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan hydrochloride liposome injection combined with Capecitabine and Lenvatinib (Experimental): Patients will receive irinotecan hydrochloride liposome injection combined with Capecitabine and Lenvatinib therapy in a 2-week treatment cycle.
  Interventions: Drug: irinotecan hydrochloride liposome injection; Drug: Capecitabine; Drug: Lenvatinib

INTERVENTIONS:
Drug: irinotecan hydrochloride liposome injection — Irinotecan hydrochloride liposome injection (70mg/m2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle.
  Other Names: duoenyi
Drug: Capecitabine — Capecitabine (850 mg/m2) will be administered orally in a 2-week treatment cycle, twice a day from day 1 to day 10 of each cycle.
  Other Names: Kapeitabin
Drug: Lenvatinib — Lenvatinib (8 mg) will be administered orally in a 2-week treatment cycle, once a day from day 1 to day 14 of each cycle
  Other Names: lunfatini

SUMMARY:
To evaluate the efficacy and safety of irinotecan hydrochloride liposome injection combined with Capecitabine and Lenvatinib for second-line treatment in Patients With advanced or metastatic biliary tract carcinoma.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of irinotecan hydrochloride liposome injection combined with Capecitabine and Lenvatinib for second-line treatment in Patients With advanced or metastatic biliary tract carcinoma.

Patients will receive irinotecan hydrochloride liposome injection combined with Capecitabine and Lenvatinib therapy in a 2-week treatment cycle.

Drug: Irinotecan hydrochloride liposome injection (70mg/m2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle.

Drug: Capecitabine (850 mg/m2) will be administered orally in a 2-week treatment cycle, twice a day from day 1 to day 10 of each cycle.

Drug: Lenvatinib (8 mg) will be administered orally in a 2-week treatment cycle, once a day from day 1 to day 14 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years
2. Has histologically confirmed diagnosis of advanced (metastatic) and/or unresectable (locally advanced) biliary tract cancer (intra-or extrahepatic cholangiocarcinoma or gallbladder cancer)
3. For subjects who have progressed after receiving previous first-line therapy, relapse within 6 months after the end of (neo) adjuvant therapy is considered as first-line therapy failure
4. The previous treatment regimen should be free of capecitabine and Lenvatinib, and the time of recurrence diagnosis should be greater than 6 months after the last dose, with no delayed toxic reactions
5. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
6. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1
7. Has a life expectancy of greater than 3 months
8. LVEF≥50%，no obvious abnormalities in myocardial enzyme spectra
9. Good bone marrow function：ANC ≥1.5×109/L, Hb≥90g/L.PLT ≥100×109/L, WBC≥3.0×109/L
10. Liver function：ALT/AST ≤ 2.5 x ULN; When there is liver metastasis, ALT/AST ≤ 5 x ULN，total bilirubin ≤1.5 x ULN
11. Renal function：Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60mL/min (according to Cockcroft-Gault formula)
12. Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT) and international standardized ratio (INR) ≤1.5×ULN
13. Urine routine results showed that urine protein <2+; For patients with urine protein ≥2+ at baseline, 24-hour urine collection and 24-hour urine protein quantification <1g should be performed.
14. Patients with biliary obstruction or no evidence of persistent infection should receive adequate biliary drainage; Active or suspected infection is not allowed
15. Adverse reactions caused by previous treatment must be restored to grade 1 or baseline according to CTCAE5.0 (except for toxicity such as alopecia, grade 2 and below peripheral neuropathy, which can be included after the investigator determines that there is no safety risk).
16. Non-pregnant or lactating female; Effective contraception should be used by female/Male of childbearing age during the study period and for 6 months after the end of study treatment
17. There were no contraindications for the use of irinotecan liposomes, capecitabine and Lenvatinib
18. The patient had good compliance, could understand the research process of this study, and signed a written informed consent

Exclusion Criteria:

1. Patients who have had other malignant tumors within the previous 5 years (except cured carcinoma in situ and skin basal cell carcinoma)
2. Uncontrolled pleural effusion or ascites
3. History of gastrointestinal bleeding or significant tendency to gastrointestinal bleeding within 6 months before the study, such as esophageal and gastric varices with bleeding risk, active local ulcers, and continuous positive fecal occult blood
4. A deep vein thrombosis or embolism event occurred within 6 months before the start of treatment
5. any known brain or meningeal metastases
6. Subjects were co-administered a potent CYP3A4 inducer within 3 weeks prior to first dosing, or a potent CYP3A4 inhibitor or a potent UGT1A1 inhibitor within 3 weeks prior to first dosing
7. Subjects underwent large organ surgery (except needle biopsy, central venous catheterization, port catheterization, stenting for relief of biliary obstruction, percutaneous hepatobiliary drainage, and cholecystostomy) or an elective surgical program within 4 weeks before the first dose of the study drug
8. Subjects had an active infection or unexplained fever >38.5 degrees during screening or before the first dose (the investigator determined that the subject's fever due to the tumor could be enrolled)
9. Subjects with congenital or acquired immune dysfunction, such as HIV infection or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA≥1000 IU/ml; Hepatitis C reference: HCV RNA≥1000 IU/ml) Chronic hepatitis B virus carriers with HBV DNA < 2000 IU/ml must also receive antiviral therapy during the trial to be enrolled
10. Subject has homozygous mutation or double heterozygous mutation of UGT1A1 allele
11. There are serious concomitant diseases: such as uncontrolled diabetes after hypoglycemic drug treatment, uncontrolled hypertension, serious cardiovascular and cerebrovascular disease, kidney failure, liver failure, uncontrolled epilepsy, central nervous system disease or mental disorder history, clear gastrointestinal bleeding tendency, intestinal paralysis, intestinal obstruction, etc
12. Grade 1 diarrhea with an increase in the number of stools > 4 times per day compared to baseline; The moderate and severe effluents from stoma increased; Limited activities of daily living with the aid of tools or even self-rational activities of daily living; Life-threatening; Need urgent medical attention
13. Had participated in other clinical investigators within 4 weeks before enrollment
14. Unsuitable for participation in the trial by the investigator assessed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
Objective response rate (ORR) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor
overall survival (OS) | baseline up to approximately 12 month
  To evaluate the efficacy of anti-tumor
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the initiation of the first dose to 14 days after the last dose
  To identify the incidence of AE and SAE in clinical trial
Time to treatment failure (TTF) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor
Quality of life (QoL) | baseline up to approximately 12 months
  To identify the quality of life by QLQ-C30 V3.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiujuan Qu, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, China